CLINICAL TRIAL: NCT05041322
Title: Improving Ventilatory Capacity in Those With Chronic High Level SCI
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Spaulding Rehabilitation Hospital (Other)
Responsible Party: Principal Investigator, J. Andrew Taylor, Ph.D., Director, Cardiovascular Research Laboratory, Spaulding Rehabilitation Hospital
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: 2016P002409
Record Dates: First submitted 2021-08-06; First posted 2021-09-13 (Actual); Results first posted 2025-09-18 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Spinal Cord Injuries
Keywords: Pulmonary Function Test; Buspirone Hydrochloride; Oxygen Consumption
MeSH Terms: conditions — Spinal Cord Injuries | interventions — Buspirone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator): Subjects take placebo pills (twice a day) for 14 Days.
  Interventions: Drug: Placebo
- Buspirone (Active Comparator): Subjects take 30 mg buspirone HCl (15 mg twice a day) for 14 Days.
  Other Names:
  Buspar
  Interventions: Drug: Buspirone

INTERVENTIONS:
Drug: Buspirone — Subjects take 30 mg buspirone HCl (15 mg twice a day) for 14 Days.
  Other Names: BuSpar, Buspirone Hydrochloride
  Arms: Buspirone
Drug: Placebo — Subjects take placebo pills (twice a day) for 14 Days.
  Other Names: Control
  Arms: Placebo

SUMMARY:
The purpose of this study is to find out if taking the drug Buspar will increase breathing capacity in individuals with spinal cord injuries.

DETAILED DESCRIPTION:
Chemoreceptive regulatory feedback is crucial for precise ventilatory control, especially during exercise. However, individuals with high-level SCI have a reduced chemoreceptive drive to breathe. Studies have shown lesser increases in minute ventilation and mouth pressure during hypercapnia in those with tetraplegia. Peripheral factors rather than central factors appear to cause the reduction of the ventilatory response to hypercapnia. This reduced ventilatory drive may have functional impact on exercise ventilation in patients with high level SCI and enhancing ventilatory drive may improve exercise ventilation in high-level SCI.

Currently, there are no treatments to overcome these functional deficits that affect daily activity and exercise-based rehabilitation recovery. However, previous work in an animal model of SCI has found that that a serotonin agonist markedly increases respiratory responses to carbon dioxide. Treatment with a serotonin 5HT1A agonist effectively improved the ventilatory drive after both acute and chronic spinal cord injuries in rats. One potential mechanism is increased excitability of the ventral motoneurons that have survived the spinal cord injury. 5-HT1A receptors do exist on these neurons, and when activated, amplify the excitatory output. Another mechanism resides at the intercostal and abdominal muscle afferents which influence supraspinal respiratory group neurons in the brainstem and motor output to the muscles of breathing. Hence, serotonin agonists may act on neural pathways in the spinal cord responsible for transferring afferent information from intercostal muscles to supraspinal centers. Lastly, 5-HT1A receptors may also be involved in functional plasticity of neural respiratory pathways, in particular ipsilateral phrenic nerve activity. Up regulation of 5-HT1A receptors due to denervation supersensitivity could result in postsynaptic hyperresponsivity due to loss of descending input.

BuSpar/Buspirone is a serotonin 5HT1A agonist and used as an anxiolytic in humans. It does not cause sedation, has minimal effects on psychomotor performance or cognition, and has low threshold for abuse potential or dependence liability. Prior studies have found Buspirone to be well tolerated. It has been used safely in spinal cord injury, but not for respiratory purposes. (Though there is one clinical trial in process: Role of Enhancing Serotonin Receptors Activity for Sleep Apnea Treatment in Patients with SCI.) However, Buspirone up to 60 mg daily has been used to treat disturbed respiratory rhythms in multiple sclerosis, brain cancer, and brainstem infarction. Interestingly, in patients with COPD, a 14-day oral administration of buspirone (20 mg) found improved anxiety and depression as well as increased exercise tolerance with lesser sensations of dyspnea. Hence, buspirone may offer a treatment to improve hypercapnic ventilatory drive. Given that oral administration of 30 mg results in peak plasma levels at one hour and that the average elimination half life is about 2 to 3 hours, buspirone is an attractive and safe approach to exploring the ability to improve respiratory responses to exercise and/or hypercapnia exposure in those with high level spinal cord injury that limits breathing capacity.

ELIGIBILITY:
Inclusion Criteria:

* Chronic high-level SCI (at least 24-months post injury)
* Age 18 to 50 years.
* Medically stable
* Spinal Cord Injury ≥T3
* American Spinal Injury Association grade A or B or C.
* Able to perform arm crank exercise.

Exclusion Criteria:

* Cardiomyopathy
* High blood pressure( >140/90 mmHg or you are taking high blood pressure medication)
* Significant irregular heartbeat
* Heart disease
* Chronic lung disease (COPD, bronchitis)
* Current use of cardioactive or antidepressant drugs
* Family history of significant irregular heart beat or sudden cardiac death
* Orthostatic hypotension (symptomatic fall in blood pressure >30 mmHg when upright)
* Current grade 2 or greater pressure ulcers at relevant contact site
* Neurological disease (stroke, peripheral neuropathy, myopathy)
* Arm or shoulder conditions that limit ability to perform arm crank exercise
* History of bleeding disorder, diabetes, kidney disease, cancer, other neurological disease
* Recent weigh change (greater than 10 pounds)
* Regular use of tobacco
* Intrathecal baclofen pump,
* Current use of cardioactive, antidepressant, other sedating agents
* Suicidal ideation
* Pregnant and/or breastfeeding women.

In addition, subjects must have no known hypersensitivity to Buspar and must not be taking a monoamine oxidase inhibitor.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2020-11-29 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2024-11-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Spaulding Hospital Cambridge, Cambridge, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Individuals with a medically stable spinal cord injury at neurological level >T3 and AIS A, B, or C were recruited 2021-22 to participate in the study.
Pre-assignment Details: Excluded if they have cardiovascular disease, diabetes, other neurological disease, renal disease, or cancer. Also excluded with current use of tobacco, cardioactive medications, antidepressants, or sedating agents.
Groups:
- Placebo Then Buspirone; Buspirone Then Placebo: If eligible, all participants were studied at baseline before being randomly assigned to a 14 days of treatment (placebo or busrpirone) before crossing over to the other arm.
Period: Baseline
Arm/Group | Placebo Then Buspirone | Buspirone Then Placebo
Started (An additional 4 individuals signed an informed consent but withdrew before randomization.) | 5 | 4
Completed | 4 | 4
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Period: Treatment 1 (14 Days)
Arm/Group | Placebo Then Buspirone | Buspirone Then Placebo
Started | 4 | 4
Completed | 2 | 3
Not Completed | 2 | 1
Not completed — Adverse Event | 1 | 0
Not completed — Withdrawal by Subject | 1 | 1
Period: Treatment 2 (14 Days)
Arm/Group | Placebo Then Buspirone | Buspirone Then Placebo
Started | 2 | 3
Completed | 2 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: 13 individuals signed the informed consent, 9 were randomized to treatment groups, 8 completed baseline measurements, and 5 completed the entire study including crossing over to the other treatment.
Groups:
- All Participants: If eligible, all participants were studied at baseline before being randomly assigned to a 14 days of treatment (placebo or busrpirone) before crossing over to the other arm.
Arm/Group | All Participants
Number analyzed (Participants) | 8
Age, Continuous [Mean (Standard Deviation); unit: Years] | 33.1 (8.54)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 7
  More than one race | 0
  Unknown or Not Reported | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 7
  Unknown or Not Reported | 0
Pulmonary Function [Mean (Standard Deviation); unit: L] — Forced expiratory volume over 1 second (FEV1).
  L | 3.15 (1.06)
Hypercapnic Ventilatory Response [Mean (Standard Deviation); unit: L /min/mmHg of CO2] — The drive to breathe with a change in carbon dioxide measured at baseline.
  L /min/mmHg of CO2 | 0.725 (0.525)
Sleep Quality [Mean (Standard Deviation); unit: apneas + hypopneas per hour] — Sleep apneas and hypopneas per hour at baseline Population: Equipment failure led to one sleep study not being recorded.
  apneas + hypopneas per hour
    number analyzed (Participants) | 7
    (all) | 2.85 (7.01)
Exercise Pulmonary Capacity [Mean (Standard Deviation); unit: ml/kg of O2] — Peak oxygen consumption during exercise measured on the arm crank at baseline. Population: One participant did not reach VO2max, so is not included.
  ml/kg of O2
    number analyzed (Participants) | 7
    (all) | 15.32 (7.01)

OUTCOME MEASURES:

1. Primary Outcome: Pulmonary Function
Description: Forced expiratory volume over 1 second (FEV1).
Time Frame: 14 Days
Measure: Mean (Standard Deviation); unit: L
Arm/Group | Placebo | Buspirone
Number analyzed (Participants) | 5 | 5
L | 3.59 (1.07) | 3.77 (1.12)

2. Primary Outcome: Hypercapnic Ventilatory Response
Description: A change in the drive to breathe with a change in carbon dioxide
Time Frame: 14 Days
Measure: Mean (Standard Deviation); unit: L /min/mmHg of CO2
Arm/Group | Placebo | Buspirone
Number analyzed (Participants) | 5 | 5
L /min/mmHg of CO2 | 0.659 (0.320) | 0.566 (0.133)

3. Primary Outcome: Sleep Quality
Description: Sleep apneas and hypopneas per hour.
Time Frame: 14 Days
Measure: Mean (Standard Deviation); unit: counts per hour
Arm/Group | Placebo | Buspirone
Number analyzed (Participants) | 5 | 5
counts per hour | 4.26 (2.11) | 6.18 (2.97)

4. Primary Outcome: Exercise Pulmonary Capacity
Description: Change in peak oxygen consumption during exercise
Time Frame: 14 Days
Measure: Mean (Standard Deviation); unit: ml/kg of O2
Arm/Group | Placebo | Buspirone
Number analyzed (Participants) | 5 | 5
ml/kg of O2 | 18.28 (8.20) | 17.69 (7.29)

ADVERSE EVENTS:
Time Frame: From enrollment to end of second treatment, up to 28 days.
Arm/Group | Buspirone | Placebo
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/6
Other Adverse Events (participants affected / at risk) | 0/5 | 1/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Buspirone (N=5) | Placebo (N=6)
Gastrointestinal distress (Gastrointestinal disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
Insufficient sample size to make any determination of efficacy.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-09-22): https://cdn.clinicaltrials.gov/large-docs/22/NCT05041322/Prot_SAP_000.pdf